CLINICAL TRIAL: NCT03766464
Title: Observational Study on Aspects Associated With Obstructive Sleep Apnea, Bruxism and Orofacial Pain
Brief Title: Aspects Associated With Obstructive Sleep Apnea, Bruxism and Orofacial Pain
Status: Completed | Type: Observational
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Noéli Boscato, PhD, Associate Professor, Federal University of Pelotas
Other Study IDs: FUPelotas1
Record Dates: First submitted 2018-11-06; First posted 2018-12-06 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Bruxism; Temporomandibular Joint Disorders; Obstructive Sleep Apnea Syndrome
Keywords: sleep bruxism; polisomnography; sleep wake disorders
MeSH Terms: conditions — Bruxism; Temporomandibular Joint Disorders; Sleep Apnea, Obstructive; Sleep Bruxism; Sleep Wake Disorders | interventions — Pain Threshold

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- with sleep bruxism, apnea and DTM: Patients who will undergo analysis of:
  Evaluation of TMD and pain sensitivity Evaluation of SB Evaluation of AB
  Interventions: Diagnostic Test: Evaluation of TMD and pain sensitivity; Diagnostic Test: Evaluation of SB; Diagnostic Test: Evaluation of AB

INTERVENTIONS:
Diagnostic Test: Evaluation of TMD and pain sensitivity — Extra and intraoral clinical examination will be performed and the Diagnostic Criteria for Temporomandibular Disorders (DC / TMD) questionnaire will be applied. Measurements shall be bilateral in the masseter, anterior temporal and tenar muscles and the arithmetic mean between three measurements will be considered the value for each side for pain sensitivity analysis with an dynamometer.
Diagnostic Test: Evaluation of SB — The presence or absence of SB will be diagnosed by Polysomnography
Diagnostic Test: Evaluation of AB — A smartphone will be used, which was developed for a momentary evaluation that allows a report of the exact moment of AB and its possible associated symptoms.

SUMMARY:
This study evaluated the influence of the sleep bruxism (SB), awake bruxism (AB) and obstructive sleep apnea syndrome (OSAS) on the signs and symptoms of temporomandibular disorders (TMD).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by partial or total obstruction of the upper airways. Bruxism is defined as a repetitive activity of the mandibular musculature characterized by the tightening or grinding of the teeth and/or by the retrusion or propulsion of the mandible, and according to their manifestation circadian is defined as sleep bruxism (SB) or wake bruxism (AB). This prospective clinical study will be performed with adults (20 to 60 years) and elderly (> 60 years) (WHO-World Health Organization) who will be undergone polysomnography (PSG) at a private medical outpatients clinic from January to December 2019 to evaluate the influence of SB, AB, and OSA on signs and symptoms of TMD. The individuals will be assessed clinically and diagnosed for TMD using the "Diagnostic Criteria for Temporomandibular Disorders", for SB and OSA using PSG, and AB using the smartphone application. Specific statistical tests will be determined after preliminary analysis of the data (α= 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 20 to 60 years) and elderly (aged > 60 years) (WHO-World Health Organization, 2015) who will be undergone PSG at the Pelotas Sleep Institute (ISP);
* Adequate cognitive capacity to understand and answer the questionnaire.

Exclusion Criteria:

• Those which the participants were unable to answer the questionnaires and who presented a history of epilepsy that could interfere in the results of PSG.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults (aged 20 to 60 years) and elderly (aged > 60 years) who had undergone PSG at the Pelotas Sleep Institute (ISP), a private medical outpatients clinic, from January to December 2019, will be invited to participate in the study. Written consent was given by all participants who agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Polisomnography analysis | 4 months after study start
  Patients included in the study will receive polisomnography exams for diagnosis of SB and OSAS. The data will be obtained from polisomnography records

SECONDARY OUTCOMES:
TMD assessment | 6 months after study start
  All patients who had undergone polisomnography will answer the DC / TMD questionaire and clinical exams.
Diagnosis of awake bruxism | 8 months after study start
  All patients will use a Smartphone application after undergone polisomnography
TMD pain | 10 months after study start
  All patients who had undergone polisomnography will answer the DC / TMD questionaire and clinical exams with algometer.

CONTACTS AND LOCATIONS:
Overall Officials: Noéli Boscato, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Noéli Boscato, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] [1] Lobbezoo F, Ahlberg J, Glaros AG, Kato T, Koyano K, Lavigne GJ, Leeuw LR, Manfredini D, Winocur, E. Bruxism defined and graded: an international consensus. J Oral Rehabil. 2013;40:2-4. [2] Lobezzo F, Naeije M. Bruxism is mainly regulated centrally, not peripherally. J Oral Rehabil. 2001;28:1085-1091. [3] Lavigne GJ, Khoury S, Abe S, Yamaguchi T, Raphael K. Bruxism physiology and pathology: an overview for clinicians. J Oral Rehabi. 2008;35:476-494. [4] Svensson P, Arima T, Lavigne G, Castrillon E. Sleep Bruxism: Definition, Prevalence, Classification, Etiology, and Consequences, In: Kryger M, Roth T, Dement WC (eds), Principles and Practice of Sleep Medicine, 7th edition, 2020, chapter 171. [5] Lobbezoo F, Ahlberg J, Raphael KG, Wetselaar P, Glaros AG, Kato T, et al. International consensus on the assessment of bruxism: Report of a work in progress. J Oral Rehabil. 2018;45:837-44. [6] American Academy of Sleep Medicine (AASM). International Classification of Sleep Disorders. 3rd ed. ed. Darien, IL: American Academy of Sleep Medicine; 2014. [7] Louca M, Short MA. The effect of one night's sleep deprivation on adolescent neurobehavioral performance. Sleep. 2014;37:1799-1807.. [8] Casett E, Réus JC, Stuginski-Barbosa J, Porporatti AL, Carra MC, Peres MA, De Luca Canto D, Manfredini, D. Validity of different tools to assess sleep bruxism: a meta-analysis. J Oral Rehabil. 2017;44:722-734. [9] Schroeder K, Gurenlian JR. Recognizing poor sleep quality factors during oral health evaluations. Clin Med Res. 2019;17: 20-28. [10] Ramzy JA, Rengan R, Mandal M, Rani S, Sanchez MV, Jaffe F, Krachman S. Hypoxic Burden and Apnea-Hypopnea Duration in Patients with Positional Obstructive Sleep Apnea. Sleep. 2020;43:A217-A218. [11] Baad-Hansen L, Thymi M, Lobbezoo F, Svensson P. To what extent is bruxism associated with musculoskeletal signs and symptoms? A systematic review. J Oral Rehabil. 2019;46:845-861. [12] Ferreira MC, Porto de Toledo I, Dutra KL, Stefani FM, Porporatti AL, Flores-Mir C, De Luca Canto G. Association between chewing dysfunctions and temporomandibular disorders: A systematic review. J Oral Rehabil. 2018;45:819-835. [13] Amorim CSM, Vieira GF, Firsoff EFO, Frutuoso JRC, Puliti E, Marques AP. Symptoms in different severity degrees of bruxism: a cross-sectional study. Fisio Pesq, 2016;23:423-430. [14] Sessle BJ, Adachi K, Yao D, Suzuki Y, Lavigne GJ. Orofacial pain and sleep. Contemp Oral Med. 2017;1-27. [15] Manfredini D, Ahlberg J, Castroflorio T, Poggio CE, Guarda-Nardini L, Lobbezoo F. Diagnostic accuracy of portable instrumental devices to measure sleep bruxism: a systematic literature review of polysomnographic studies. J Oral Rehabil. 2014;41:836-842. [16] Wetselaar P, Vermaire E, Lobbezoo F, Schuller AA. The prevalence of awake bruxism and sleep bruxism in the Dutch adult population. J Oral Rehabi. 2019;46:617-623. [17] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP, et al. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014;12:1495-9. [18] World Health Organization (WHO). Obesity and overweight. Fact sheet 2016